CLINICAL TRIAL: NCT03922113
Title: Muscle Strength and Function After Intensive Care, Compared to Surgical and Healthy Subjects
Brief Title: Muscle Function After Intensive Care
Status: Completed | Type: Observational
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Rousseau, Head of Clinic, University of Liege
Other Study IDs: FAIC
Record Dates: First submitted 2019-04-13; First posted 2019-04-19 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Critically Ill; Colorectal Surgery; Healthy; Muscle Strength
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Critically ill patients: Patients who spent a minimum of 48h in ICU
  Interventions: Other: Patient follow up
- Surgical patients: Patients who were scheduled for elective colorectal surgery
  Interventions: Other: Patient follow up
- Healthy subjects: Healthy volunteers
  Interventions: Other: Patient follow up

INTERVENTIONS:
Other: Patient follow up — Patient follow up during one month

SUMMARY:
Final objective of critical care is no longer only survival. The role of medical and paramedical teams should also be to restore functional capacities, autonomy and quality of life. What has been call "intensive care unit - acquired weakness" (ICU-AW) is associated to acute and long term increased mortality, prolonged ICU and hospital stay, prolonged duration of mechanical ventilation, altered quality of life in survivors and increased health-related costs. In order to target efficient secondary prevention and early rehabilitation, prompt identification of muscle weakness is crucial. Several methods, aiming to assess muscle mass, muscle strength or physical function, are described. Manual muscle testing using the Medical Research Council (MRC) scale is still the most commonly utilized tool to diagnose ICU-AW (MRC <48/60). Dynamometry is an objective alternative and one of the most accurate clinimetric tool to assess muscle strength. Literature is overflowing with insufficiently standardized dynamometry data. Using the investigator's published standardized protocol of quadriceps strength (QS) assessment, this observational study aim to describe physical performances of CC patients and thus to define the weakest ones, by comparing them to surgical and healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Collaborative ICU patients with length of stay > 48h
* Surgical patients scheduled for colorectal surgery
* Healthy subjects

Exclusion Criteria:

* a score > 1 or < -1 on the Richmond Agitation and Sedation Scale (RASS)
* coma
* total hip or knee arthroplasty in the dominant limb
* unauthorized support on the dominant leg
* open wound located at the ankle's anterior face of the dominant leg
* pre-existing myopathy or polyneuropathy
* para- or tetraparesis, para- or tetraplegia
* refusal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Collaborative ICU patients with length of stay > 48h
  * Surgical patients scheduled for colorectal surgery
  * Healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Change in Quadriceps strength | For critically ill patients: T0 (as soon as they were collaborative in ICU) and M1 (at one month following discharge), for surgical patients at T0 (day before surgery) and at M1 (one month following discharge), for healthy subjects: T0
  Maximal isometric voluntary quadriceps contraction is assessed using a hand-held dynamometer (MicroFet2®, Hoggan Health Industries, West Jordan, UT, USA) with a curved transducer pad. The highly standardized protocol is detailed in a previously published validation study (Rousseau et al, Acta Anaesthesiologica Belgica 2018). Measurements are performed at bedside with patient lying on supine position. The dominant limb is tested (kicking leg). The best performance out of 3 measurements is considered for the analysis. Muscle strength is expressed in Newton (N). Relative strength, normalized according to actual body weight, is expressed in N/kg.

SECONDARY OUTCOMES:
Change in Medical Research Council test (MRC) | For critically ill patients: T0 (as soon as they were collaborative in ICU) and M1 (at one month following discharge), for surgical patients at T0 (day before surgery) and at M1 (one month following discharge), for healthy subjects: T0
  Manual evaluation of muscle strength. This scale grades muscle power on a scale of 0 to 5 in relation to the maximum expected for that muscle. Grade 0 = no movement is observed, grade 5= muscle contracts normally against full resistance. Six muscles groups are tested at both sides of the body: shoulder abduction, elbow flexion, wrist extension, hip flexion, knee extension, ankle dorsiflexion. Maximal total score is 60.
Change in 4-items Physical Function Intensive care Test (PFIT-s) | For critically ill patients: T0 (as soon as they were collaborative in ICU) and M1 (at one month following discharge), for surgical patients at T0 (day before surgery) and at M1 (one month following discharge), for healthy subjects: T0
  This test measures strength and functional outcomes, by ranking 4 components: assistance (sit and stand), cadence (steps/min), shoulder flexion strength and knee extension strength. Maximal score is 10.
Change in Barthel index for activities of daily living | For critically ill patients: T0 (as soon as they were collaborative in ICU) and M1 (at one month following discharge), for surgical patients at T0 (day before surgery) and at M1 (one month following discharge), for healthy subjects: T0
  This score assesses functional independence by ranking patient's independence in the following areas: feeding, bathing, grooming, dressing, bowel control, bladder control, toilet use, transfers, mobility in level surfaces and stairs. Maximal total score is 100 = totally independent).

IPD SHARING:
Plan to Share IPD: No